CLINICAL TRIAL: NCT05517174
Title: A Pragmatic Randomized Trial to Evaluate the Effectiveness of High-Dose Quadrivalent Influenza Vaccine vs. Standard-Dose Quadrivalent Influenza Vaccine in Older Adults
Acronym: DANFLU-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Collaborators: Sanofi (Industry); Statens Serum Institut (Other)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, PhD, MPH, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DANFLU-2; 2022-500657-17-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2022-08-20; First posted 2022-08-26 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Influenza
Keywords: Influenza; Vaccination; Pragmatic; Registry; Pneumonia; Respiratory; Cardiovascular
MeSH Terms: conditions — Influenza, Human; Pneumonia | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Dose Quadrivalent Influenza Vaccine (Experimental): QIV-HD single injection at Day 0
  Interventions: Biological: High-Dose Quadrivalent Influenza Vaccine
- Standard-Dose Quadrivalent Influenza Vaccine (Active Comparator): QIV-SD single injection at Day 0
  Interventions: Biological: Standard-Dose Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: High-Dose Quadrivalent Influenza Vaccine — For this arm, the high-dose quadrivalent influenza vaccine Efluelda®/Fluzone® High-Dose Quadrivalent will be used.
  Other Names: QIV-HD
  Arms: High-Dose Quadrivalent Influenza Vaccine
Biological: Standard-Dose Quadrivalent Influenza Vaccine — Any standard-dose quadrivalent influenza vaccine administered in the Danish governmental influenza vaccine program may be used.
  Other Names: QIV-SD
  Arms: Standard-Dose Quadrivalent Influenza Vaccine

SUMMARY:
The purpose of this pragmatic randomized trial is to evaluate the relative vaccine effectiveness of high-dose quadrivalent influenza vaccine (QIV-HD) vs. standard-dose quadrivalent influenza vaccine (QIV-SD) in older adults. Participants will be randomized 1:1 to either QIV-HD or QIV-SD.

DETAILED DESCRIPTION:
The study is a pragmatic, registry-based, open-label, active-controlled, individually randomized trial. The Danish nationwide administrative health registries will be used for data collection including baseline information, follow-up data, and safety monitoring. The study aims to randomize 339,700 participants over 3 influenza seasons. In each season, participants will be individually randomized 1:1 to receive either QIV-HD or QIV-SD. During the 2023/2024 and 2024/2025 seasons, up to 12,000 participants will be enrolled in a sub-cohort where participants are asked to perform home self-swabs and answer symptom questionnaires in case of influenza-like illness to enable further assessment of the impact of QIV-HD vs. QIV-SD on patient-reported outcomes among individuals with influenza-like illness and laboratory-confirmed influenza.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and above (this inclusion criterion will be modified according to the Danish government's official recommendations for the 2022/2023 and 2023/2024 influenza seasons)
* Informed consent form has been signed and dated

Exclusion Criteria:

* There are no specific exclusion criteria for this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 332438 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Hospitalization for influenza or pneumonia | ≥14 days after vaccination up to 8 months

SECONDARY OUTCOMES:
Hospitalization for any cardio-respiratory disease | ≥14 days after vaccination up to 8 months
All-cause hospitalization | ≥14 days after vaccination up to 8 months
All-cause mortality | ≥14 days after vaccination up to 8 months
Hospitalization for influenza | ≥14 days after vaccination up to 8 months
Hospitalization for pneumonia | ≥14 days after vaccination up to 8 months

OTHER OUTCOMES:
Hospitalization for influenza or pneumonia (alternate definition) | ≥14 days after vaccination up to 8 months
Hospitalization for pneumonia (alternate definition) | ≥14 days after vaccination up to 8 months
Hospitalization for influenza (alternate definition) | ≥14 days after vaccination up to 8 months
Hospitalization for any respiratory disease | ≥14 days after vaccination up to 8 months
Hospitalization for any cardiovascular disease | ≥14 days after vaccination up to 8 months
Hospitalization for myocardial infarction | ≥14 days after vaccination up to 8 months
Hospitalization for heart failure | ≥14 days after vaccination up to 8 months
Hospitalization for atrial fibrillation | ≥14 days after vaccination up to 8 months
Hospitalization for stroke | ≥14 days after vaccination up to 8 months
Major adverse cardiovascular events (MACE) defined as a composite of hospitalization for acute myocardial infarction, hospitalization for stroke, and cardiovascular death | ≥14 days after vaccination up to 8 months
MACE defined as a composite of hospitalization for acute myocardial infarction, hospitalization for stroke, hospitalization for heart failure, and cardiovascular death (alternate definition #1) | ≥14 days after vaccination up to 8 months
MACE defined as a composite of hospitalization for acute myocardial infarction, hospitalization for stroke, and all-cause death (alternate definition #2) | ≥14 days after vaccination up to 8 months
Hospitalization requiring mechanical ventilation | ≥14 days after vaccination up to 8 months
Laboratory-confirmed influenza | ≥14 days after vaccination up to 8 months
Laboratory-confirmed pneumococcal pneumonia | ≥14 days after vaccination up to 8 months
Laboratory-confirmed COVID-19 | ≥14 days after vaccination up to 8 months
Cardio-respiratory mortality | ≥14 days after vaccination up to 8 months
Respiratory mortality | ≥14 days after vaccination up to 8 months
Cardiovascular mortality | ≥14 days after vaccination up to 8 months
In-hospital mortality | ≥14 days after vaccination up to 8 months
Intensive care unit admission | ≥14 days after vaccination up to 8 months
Laboratory-confirmed influenza hospitalization | ≥14 days after vaccination up to 8 months
Any hospital contact associated with laboratory-confirmed influenza | ≥14 days after vaccination up to 8 months
Any exacerbation of pre-existing chronic obstructive pulmonary disease | ≥14 days after vaccination up to 8 months
Any exacerbation of pre-existing chronic obstructive pulmonary disease (alternate definition) | ≥14 days after vaccination up to 8 months
Severe exacerbation of pre-existing chronic obstructive pulmonary disease | ≥14 days after vaccination up to 8 months
Severe exacerbation of pre-existing chronic obstructive pulmonary disease (alternate definition) | ≥14 days after vaccination up to 8 months
Any exacerbation of pre-existing asthma | ≥14 days after vaccination up to 8 months
Any exacerbation of pre-existing asthma (alternate definition) | ≥14 days after vaccination up to 8 months
Severe exacerbation of pre-existing asthma | ≥14 days after vaccination up to 8 months
Severe exacerbation of pre-existing asthma (alternate definition) | ≥14 days after vaccination up to 8 months
Exacerbation of pre-existing heart failure | ≥14 days after vaccination up to 8 months
Exacerbation of pre-existing heart failure (alternate definition) | ≥14 days after vaccination up to 8 months
Hospitalization for pericarditis | ≥14 days after vaccination up to 8 months
Hospitalization for myocarditis | ≥14 days after vaccination up to 8 months
New-onset dementia | ≥14 days after vaccination up to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, PhD, MPH, Study Chair — Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte
Locations (2):
- Denmark (2):
  - Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup, Capital Region
  - Danske Lægers Vaccinations Service, Søborg

IPD SHARING:
Plan to Share IPD: Yes
In this trial, baseline and endpoint data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor-investigator in case of any inquiries.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Nielsen AB, Johansen ND, Modin D, Loiacono MM, Harris RC, Dufournet M, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Claggett BL, Janstrup KH, Bartholdy KV, Bernholm KF, Borchsenius JIH, Davidovski FS, Davodian LW, Dons M, Duus LS, Espersen C, Fussing FH, Jensen AMR, Landler NE, Langhoff ACF, Lassen MCH, Ottosen CI, Sengelov M, Skaarup KG, Pareek M, Muller-Wieland D, Solomon SD, Landray MJ, Gislason GH, Kober L, Sivapalan P, Martel CJ, Jensen JUS, Biering-Sorensen T. High-Dose vs Standard-Dose Influenza Vaccine in Older Adults With Diabetes: A Secondary Analysis of the DANFLU-2 Randomized Clinical Trial. JAMA Intern Med. 2026 Jan 12. doi: 10.1001/jamainternmed.2025.7286. Online ahead of print. PMID 41525066
- [Derived] Johansen ND, Modin D, Loiacono MM, Harris RC, Dufournet M, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Claggett BL, Janstrup KH, Bartholdy KV, Bernholm KF, Borchsenius JIH, Davidovski FS, Davodian LW, Dons M, Duus LS, Espersen C, Fussing FH, Jensen AMR, Landler NE, Langhoff ACF, Lassen MCH, Nielsen AB, Ottosen CI, Sengelov M, Skaarup KG, Solomon SD, Landray MJ, Gislason GH, Kober L, Ralfkiaer L, Nealon J, Sivapalan P, Martel CJ, Jensen JUS, Biering-Sorensen T. High-Dose Influenza Vaccine Effectiveness against Hospitalization in Older Adults. N Engl J Med. 2025 Dec 11;393(23):2291-2302. doi: 10.1056/NEJMoa2509907. Epub 2025 Aug 30. PMID 40888720
- [Derived] Johansen ND, Modin D, Loiacono MM, Harris RC, Dufournet M, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Claggett BL, Janstrup KH, Bartholdy KV, Bernholm KF, Borchsenius JIH, Davidovski FS, Davodian LW, Dons M, Duus LS, Espersen C, Fussing FH, Jensen AMR, Landler NE, Langhoff ACF, Lassen MCH, Nielsen AB, Ottosen CI, Sengelov M, Skaarup KG, Pareek M, Solomon SD, Landray MJ, Gislason GH, Kober L, Sivapalan P, Martel CJ, Jensen JUS, Biering-Sorensen T. High-Dose vs Standard-Dose Influenza Vaccine and Cardiovascular Outcomes in Older Adults: A Prespecified Secondary Analysis of the DANFLU-2 Randomized Clinical Trial. JAMA Cardiol. 2025 Nov 1;10(11):1186-1194. doi: 10.1001/jamacardio.2025.3460. PMID 40884442
- [Derived] Skaarup KG, Johansen ND, Modin D, Loiacono MM, Harris RC, Dufournet M, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Claggett BL, Bartholdy KV, Bernholm KF, Borchsenius JIH, Davidovski FS, Davodian LW, Dons M, Duus LS, Espersen C, Fussing FH, Jensen AMR, Landler NE, Langhoff ACF, Lassen MCH, Nielsen AB, Ottosen CI, Sengelov M, Solomon SD, Landray MJ, Gislason GH, Kober L, Sivapalan P, Martel CJ, Jensen JUS, Mebazaa A, Biering-Sorensen T. High-Dose Versus Standard-Dose Influenza Vaccine in Heart Failure: A Prespecified Analysis of the DANFLU-2 Trial. Circ Heart Fail. 2025 Nov;18(11):e013678. doi: 10.1161/CIRCHEARTFAILURE.125.013678. Epub 2025 Aug 30. PMID 40884411
- [Derived] Davidovski FS, Skaarup KG, Johansen ND, Modin D, Shaikh N, Bartelt-Hofer J, Loiacono MM, Harris RC, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Jessen R, Steenhard N, Claggett BL, Solomon SD, Kober L, Sivapalan P, Jensen JUS, Martel CJ, Biering-Sorensen T. Patient-reported outcomes and home-based self-swabs for influenza-like illness events - lessons learned from the 2023/2024 DANFLU-2 Homeswab PRO substudy. J Patient Rep Outcomes. 2025 Aug 22;9(1):108. doi: 10.1186/s41687-025-00936-8. PMID 40844659
- [Derived] Johansen ND, Modin D, Loiacono MM, Harris RC, Dufournet M, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Claggett BL, Skaarup KG, Davidovski FS, Solomon SD, Landray MJ, Gislason GH, Kober L, Sivapalan P, Martel CJ, Jensen JUS, Biering-Sorensen T. A pragmatic individually randomized trial to evaluate the effectiveness of high-dose vs standard-dose influenza vaccine in older adults: Rationale and design of the DANFLU-2 trial. Am Heart J. 2026 Jan;291:186-198. doi: 10.1016/j.ahj.2025.07.069. Epub 2025 Jul 30. PMID 40749884